CLINICAL TRIAL: NCT03313687
Title: SafeTy and Outcome of contemPorary Treatment Strategies for Cardiogenic SHOCK - an International, Observational Registry
Brief Title: SafeTy and Outcome of contemPorary Treatment Strategies for Cardiogenic SHOCK
Acronym: STOP-SHOCK
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, PD Dr. Dirk Westermann, Professor, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: STOP-SHOCK
Record Dates: First submitted 2017-10-14; First posted 2017-10-18 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
International, observational registry to investigate the outcome in patients with cardiogenic shock. The primary aim of this study is to investigate the clinical outcome of patients in cardiogenic shock.

DETAILED DESCRIPTION:
There is a focus on interventional therapies, mechanical circulatory support and new cardiovascular therapeutics in patients with cardiogenic shock (CS). The investigators will describe current practice in study sites including concomitant patients with CS. Therefore, the investigators will monitor drug therapies initiated, devices being utilized as well as outcome and side effect of possible interventions

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiogenic shock treated at a tertiary care hospital.

Exclusion Criteria:

* Age ≤17 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a tertiary care hospital.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Within 30 days after admission.
  by registration office

SECONDARY OUTCOMES:
Ischemic events, bleeding events, heart failure, sepsis, dialysis. | Within 30 days after admission.
  by survey, number of ischemic events, number of bleeding events, number of patients developing heart failure as well as heart failure severity (NYHA), patients developing terminal kidney failure requiring dialysis.
All-cause mortality | Within 12 months after admission.
  by registration office
Ischemic events, bleeding events, heart failure, sepsis, dialysis. | Within 12 months after admission.
  by survey, number of ischemic events, number of bleeding events, number of patients developing heart failure as well as heart failure severity (NYHA), patients developing terminal kidney failure requiring dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Westermann, MD, Principal Investigator — UHZ
Locations (1):
- University Heart Center, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schrage B, Ibrahim K, Loehn T, Werner N, Sinning JM, Pappalardo F, Pieri M, Skurk C, Lauten A, Landmesser U, Westenfeld R, Horn P, Pauschinger M, Eckner D, Twerenbold R, Nordbeck P, Salinger T, Abel P, Empen K, Busch MC, Felix SB, Sieweke JT, Moller JE, Pareek N, Hill J, MacCarthy P, Bergmann MW, Henriques JPS, Mobius-Winkler S, Schulze PC, Ouarrak T, Zeymer U, Schneider S, Blankenberg S, Thiele H, Schafer A, Westermann D. Impella Support for Acute Myocardial Infarction Complicated by Cardiogenic Shock. Circulation. 2019 Mar 5;139(10):1249-1258. doi: 10.1161/CIRCULATIONAHA.118.036614. PMID 30586755